CLINICAL TRIAL: NCT04793568
Title: Human Recombinant Interferon Gamma-1b for the Prevention of Hospital-acquired Pneumonia in Critically Ill Patients: a Double-blind, International, Phase 2, Randomized, Placebo-controlled Trial - the PREV-HAP Study
Acronym: PREV-HAP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RC20_0082
Record Dates: First submitted 2021-02-24; First posted 2021-03-11 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Critically Ill Patients

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recombinant Interferon gamma 1b (IMUKIN®) (Experimental)
  Interventions: Drug: Recombinant Interferon gamma 1b (IMUKIN®)
- Recombinant Interferon gamma 1b placebo (Placebo Comparator)
  Interventions: Drug: Recombinant Interferon gamma 1b placebo

INTERVENTIONS:
Drug: Recombinant Interferon gamma 1b (IMUKIN®) — 100 µg/0,5ml subcutaneous injections from day 1 to day 9 (5 injections, i.e. 1 injection of 100 µg every 48h)
  Arms: Recombinant Interferon gamma 1b (IMUKIN®)
Drug: Recombinant Interferon gamma 1b placebo — 5 subcutaneous injections from day 1 to day 9 (i.e. 1 injection of 0,5ml every 48h).
  Arms: Recombinant Interferon gamma 1b placebo

SUMMARY:
PREV-HAP study is part of a larger project entitled 'Host-targeted Approaches for the Prevention and the treatment of Hospital-Acquired Pneumonia' (HAP2), funded by the European Union's H2020 research and innovation programme under grant agreement N°847782. HAP2 aims to develop stratified host-directed drugs and biomarkers to enhance the prevention and the treatment of HAP and develop precision medicine in infectious diseases. Its ambition is to revolutionize the management of HAP: capitalising on the novel concept of critical-illness related immunosuppression altering the host-pathogens interactions, the aim is to propose a complete reappraisal of the physiopathology of HAP based on the concept of respiratory dysbiosis.

The main hypothesis of the PREV-HAP study is that human recombinant Interferon gamma 1b (rHuIFN-γ, Imukin) treatment can restore immunity in critically ill patients and prevent Hospital-Acquired Pneumonia.

The hypothesesis is that the in vivo investigations of the host-pathogens interactions can be used for the stratification of patients into high/low risk and responders/non-responders to host-targeted prevention of hospital-acquired infections.

The involvement of a state of critical-illness related immunosuppression in the susceptibility to hospital-acquired pneumonia is widely accepted, and an emerging trend is that the development of drugs for the treatment of this acquired immunosuppression will prevent infection and enhance outcomes of hospitalized patients.

It has been demonstrated that the productions of IFN-γ by immune cells are decreased in critically ill patients, and that these defects are associated with the susceptibility to HAP. rHuIFN-γ has neither been tested nor is recommended as adjunctive treatment of patients with HAP. Based on these specific factors identified in the host response, it is proposed in this study to use rHuIFN-γ as novel preventive approach for HAP.

DETAILED DESCRIPTION:
200 adult patients hospitalized in intensive care units, under mechanical ventilation in three European countries will be included in the trial, and will be randomized in 2 arms :

Arm 1 (rHu-IFNγ):

• Recombinant Interferon gamma 1b (IMUKIN®, from Clinigen®): 100 µg/0,5ml subcutaneous injections from day 1 to day 9 (5 injections, i.e. 1 injection of 100 µg every 48h),

Arm 2 (Placebo):

• Recombinant Interferon gamma 1b placebo: 5 subcutaneous injections from day 1 to day 9 (i.e. 1 injection of 0,5ml every 48h).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18yr to 85yr).
* Hospitalized in intensive care unit for less than 48 hours.
* Receiving invasive mechanical ventilation at the time of inclusion.
* One or more acute organ failure at the time of inclusion among: neurological (Glasgow coma scale <13 before sedation), hemodynamic (norepinephrine, epinephrine, or any other vasopressor at a dose of ≥ 0.1 μg per kilogram of body weight per minute or ≥0.5 mg per hour for at least 6 hours), respiratory (PaO2 / FiO2< 200) and/or renal (creatininemia > 2 fold higher than the basal value and/or oliguria < 0.5 mL/kg/hour for at less 12 hours).
* Informed consent from a legal representative, or emergency procedure (when possible according to national regulation, see below). As is not possible to obtain the patient consent prior the inclusion (comatose patients), patient consent for the study continuation will be obtained as soon as deemed possible.
* Person insured under a health insurance scheme.

Exclusion Criteria:

* Pregnant women (serum or urine test), breastfeeding women
* Patient under legal protection (incl. under guardianship or trusteeship)
* Hypersensitivity to the active substance (interferon gamma-1b) or known hypersensitivity to related products, such as another interferon, or to any of the following excipients: Mannitol, Disodium succinate hexahydrate, Succinic acid, Polysorbate 20
* Severe hepatic insufficiency ( Child Pugh score B or C)
* Liver cytolysis with hepatic enzymes (AST and/or ALT) > 5N
* Severe chronic renal insufficiency (MDRD Creatinine Clearance < 10 ml/min/1.73m2)
* Immunosuppression (hematologic cancer, aplasia, chemotherapy/radiotherapy for cancer within 3 months prior to the inclusion, known infection Human immunodeficiency virus, concomitant use of any anti-graft rejection drug).
* Coma after resuscitated cardiac arrest
* Cervical spinal cord injury
* Participation to a drug interventional study within 1 month prior to the inclusion
* Hospital-acquired pneumonia before inclusion in the study during the current hospitalization.
* Sustained hyperlactatemia > 5 mmol/L.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2021-11-07 (Actual); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
To demonstrate the efficiency of rHuIFN-γ for the prevention of hospital-acquired pneumonia | Day 28
  Rate of the composite outcome at day 28 made of at least one item among the following: all cause mortality and/or hospital-acquired pneumonia

SECONDARY OUTCOMES:
All-cause mortality [efficiency of rHu-IFN-γ, on pneumonia-associated morbidity and mortality reduction] | Day 28 and Day 90
  Rate of all-cause mortality at D28 and D90
Rate of HAP [efficiency] | Day 28
  Rate of HAP at D28
Bacterial ecology of the 1st episode of HAP [efficiency] | Day 28
  Bacterial ecology of the 1st episode of HAP (respiratory fluids)
Rate of ventilator-associated tracheobronchitis [efficiency] | Day 28
  Rate of ventilator-associated tracheobronchitis at D28 defined as at least two of the following criteria: body temperature >38°C; leukocytosis>12000 cells/mL, leucopenia <4000 cells/mL, or purulent pulmonary secretions and a positive culture of a respiratory tract samples, without appearance of a new infiltrate or change in an existing infiltrate on chest radiography
Occurence of Acute Respiratory Distress Syndrome [efficiency] | Day 28
  Acute Respiratory Distress Syndrome within 28 days after randomization
Duration of antimicrobial therapy [efficiency] | Day 28
  Duration of antimicrobial therapy at D28, antibiotic free days at D28
Duration of mechanical ventilation [efficiency] | Day 90
  Duration of mechanical ventilation at D90, mechanical ventilation free days at D90
Duration of ICU hospitalization [efficiency] | Day 90
  Duration of ICU hospitalization at D90, Duration of hospitalization at D90.
Rate of SAEs and SUSARs [tolerance] | Day 15
  Rate of serious adverse effects and suspected unexpected serious adverse reaction (SUSAR) at D15
Rate of leukocytosis [tolerance] | Day 15
  Rate of leukocytosis at D15.
Rate of neutropenia [tolerance] | Day 15
  Rate of neutropenia at D15.
Rate of lymphopenia [tolerance] | Day 15
  Rate of lymphopenia at D15.
Rate of thrombopenia [tolerance] | Day 15
  Rate of thrombopenia at D15.
Rate of liver cytolysis [tolerance] | Day 15
  Rate of liver cytolysis (Increases in AST and/or ALT) at D15.
Rate of pancreatitis [tolerance] | Day 15
  Rate of pancreatitis (Increase in Lipase) at D15.
Rate of patients with episode of fever [tolerance] | Day 15
  Rate of patients with episode of fever (T° > 38.3°C)
Rate of patients with episode of headache [tolerance] | Day 15
  Rate of patients with episode of headache
Rate of patients with episode of nausea [tolerance] | Day 15
  Rate of patients with episode of nausea
Rate of allergic reaction [tolerance] | Day 15
  Rate of major allergic reaction at D15 defined as systemic epidermic reaction, anaphylactic
Incidence of injection site reaction [tolerance] | Day 15
  Occurence of injection site reaction at D15
Rate of myalgia [tolerance] | Day 15
  Rate of myalgia at D15
Rate of arthralgia [tolerance] | Day 15
  Rate of arthralgia at D15
Rate of back pain [tolerance] | Day 15
  Rate of back pain at D15
Economic efficiency of rHu-IFN-γ in the prevention of pneumonia | Day 90
  Economic endpoint at 3 months: Incremental cost effectiveness ratio (ICER). Analysis using QALYs (Quality-Adjusted Life-Years) as a measure of effectiveness. QALYs are a measure of effectiveness specifically designed for economic evaluations.
To determine the suitability of rHu-IFN-γ from the patients' and relatives' perspectives using The Short Form (36) Health Survey | Day 90
  Changes in health-related quality of life (HRQoL) from one (M1) to three months (M3) after randomization measured with the Short Form (SF)-36 scale validated in French, Greek, and Spanish he SF-36 is a 36-item self-report questionnaire with 8 domains = Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role Emotional, and Mental Health).The scores of each domain range from 0 to 100, a higher score indicating a better HRQoL.
To determine the suitability of rHu-IFN-γ from the patients' and relatives' perspectives using the Hospital Anxiety and Depression scale (HADS) | Day 90
  Changes in anxiety and depression from M1 to M3 measured with the HADS scale validated in French, Greek, and Spanish. The HADS is a 14-item self-report questionnaire with 2 domains (anxietyand depression).
  The scores for anxiety and depression range from 0 (no symptoms) to 21 (significant number of symptoms).
To determine the suitability of rHu-IFN-γ from the patients' and relatives' perspectives using Satisfaction With Life Scale (SWLS) | Day 90
  Changes in subjective well-being from M1 to M3 measured with the Satisfaction With Life Scale (SWLS) validated in French, Greek, and Spanish. The SWLS is a 5-item self-report questionnaire. The response scores to the five items are added together to provide a total score ranging from 5 (worst satisfaction level) to 35 (best level).
To determine the acceptability of rHu-IFN-γ from the patients' and relatives' perspectives | Day 90
  Adaptation of the patients to their health state and its evolution from M1 to M3 using differential item functioning and response shift analyses for HRQoL, anxiety and depression. Change in the meaning of patients' self-evaluation between groups (DIF) and over time (response shift) will be inferred by the change in the items' parameters of the Partial Credit Models.

CONTACTS AND LOCATIONS:
Locations (18):
- France (7):
  - Angers University Hospital, Angers
  - Argenteuil Hospital, Argenteuil
  - Brest University Hospital, Brest
  - Beaujon University Hospital, Clichy
  - Limoges University Hospital, Limoges
  - Nantes University Hospital, Nantes
  - Rennes University Hospital, Rennes
- Greece (6):
  - Aghioi Anargyroi General Oncology Hospital, Athens
  - Attikon University General Hospital, Athens
  - General University Hospital of Heraklion, Heraklion
  - University General Hospital of Ioannina, Ioannina
  - General University Hospital of Larissa, Larissa
  - Koutlimbaneio & Triantafylleio General Hospital of Larissa, Larissa
- Spain (5):
  - Hospital Clínic Barcelona, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hôpital universitaire Arnau de Vilanova, Lleida
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario de Son Llátzer, Palma

REFERENCES:
- [Derived] Anani H, Destras G, Regue H, Bulteau S, Bressollette-Bodin C, Roquilly A, Josset L. Metagenome-assembled complete genome of Bohxovirus, a virulent bacteriophage involved in the prediction of hospital-acquired pneumonia in intubated critically ill patients. Microbiol Resour Announc. 2025 Dec 11;14(12):e0059225. doi: 10.1128/mra.00592-25. Epub 2025 Oct 29. PMID 41159973
- [Derived] Bulteau S, Braud M, Petrier M, Castain L, Anani H, Peltier C, Mobuchon L, Bouras M, Flattres D, Poschmann J, Josset L, Roquilly A, Bressollette-Bodin C. Interferon Gamma Injection and Its Effect on the Respiratory Anelloviridae Population in ICU Ventilated Patients. J Med Virol. 2025 Oct;97(10):e70612. doi: 10.1002/jmv.70612. PMID 41036698
- [Derived] Anani H, Destras G, Bulteau S, Castain L, Semanas Q, Burfin G, Petrier M, Martin FP, Poulain C, Dickson RP, Bressollette-Bodin C, Roquilly A, Josset L. Lung virome convergence precedes hospital-acquired pneumonia in intubated critically ill patients. Cell Rep Med. 2025 Sep 16;6(9):102289. doi: 10.1016/j.xcrm.2025.102289. Epub 2025 Sep 5. PMID 40914165
- [Derived] Bouras M, Tessier P, Poulain C, Schirr-Bonnans S, Roquilly A. Three-month outcomes and cost-effectiveness of interferon gamma-1b in critically ill patients: a secondary analysis of the PREV-HAP trial. J Intensive Care. 2024 Oct 11;12(1):40. doi: 10.1186/s40560-024-00753-z. PMID 39394183